CLINICAL TRIAL: NCT04632225
Title: A Phase 2a, Double-Blind, Randomized, Placebo-Controlled, Multicenter Study to Assess the Safety of Engensis in Participants With Amyotrophic Lateral Sclerosis
Brief Title: Safety of Engensis in Participants With Amyotrophic Lateral Sclerosis
Acronym: REViVALS-1A
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Helixmith Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VMALS-002-2
Record Dates: First submitted 2020-10-29; First posted 2020-11-17 (Actual); Results first posted 2025-05-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-08

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Engensis (Active Comparator): 64 mg Engensis per Treatment Cycle, with each of 3 cycles composed of 2 days of 128 injections each to the right and left target muscles, spaced 2 weeks apart
  Interventions: Biological: Engensis
- Placebo (Placebo Comparator): 32 mL of Placebo per Treatment Cycle, with each of 3 cycles composed of 2 days of 128 injections each to the right and left target muscles, spaced 2 weeks apart
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Engensis — Lyophilized biologic to be reconstituted containing Engensis
  Arms: Engensis
Other: Placebo — Injectable liquid
  Arms: Placebo

SUMMARY:
The purpose of this study was to evaluate the safety of intramuscular administration of Engensis in Participants with Amyotrophic Lateral Sclerosis as compared to Placebo. Safety will be assessed by incidences of treatment-emergent adverse events, treatment-emergent serious adverse events, injection site reactions and other adverse events of special interest, and the clinically significant laboratory values after injections of Engensis compared to Placebo. Exploratory endpoints include assessment of muscle function using the Revised Amyotrophic Lateral Sclerosis Functional Rating Scale subscores for Fine and Gross Motor Function; muscle strength by quantitative testing using handheld dynamometry and the Accurate Test of Limb Isometric Strength where available; quality of life using the Amyotrophic Lateral Sclerosis Assessment Questionnaire-40; patient global impression of change, clinical global impression of change, and clinical global impression of severity; and evaluation of lung function using Slow Vital Capacity. Muscle biopsies will be performed during the study for future biomarker analyses.

DETAILED DESCRIPTION:
VMALS-002-2 was a controlled study to evaluate the safety of intramuscular administration of Engensis to subjects with Amyotrophic Lateral Sclerosis, as compared to Placebo. Subjects randomly assigned to Engensis were to receive a total dose of 192 mg Engensis divided into 3 treatment cycles of 64 mg Engensis each. A dosing schedule developed from those used in the Phase 1/2 Amyotrophic Lateral Sclerosis study and in three diabetic peripheral neuropathy studies were used in this study. The intramuscular injections to each target muscle group were divided into three Injection Visits (equal halves), two weeks apart on Days 0, and 14, with retreatment at Days 60 and 74, and Days 120 and 134. Engensis was delivered in a solution of 0.5 mg VM202/mL.

Results from this Phase 1/2 study suggest that targeted delivery of hepatic growth factor to motor neurons via intramuscular injections of Engensis was safe and well tolerated, based on data from 18 enrolled subjects who were followed through 90 days after the first injection [Sufit et al., 2017]. Following injections until Day 90, a plateau or a relative slowing in decline of the Amyotrophic Lateral Sclerosis Functional Rating Scale scores and muscle strength was noted, suggesting a slowing of disease progression. After 90 days, the plateau was no longer observed in the Amyotrophic Lateral Sclerosis Functional Rating Scale, with the notable exception of a trend toward better preservation of bulbar and breathing functions as measured by the Amyotrophic Lateral Sclerosis Functional Rating Scale subscore, which appeared to persist out to 180 days. The change in Amyotrophic Lateral Sclerosis Functional Rating Scale total score over time or "slope" (>0, indicating clinical stability or improvement) following Engensis treatment was greatest at 2 months in 50% of subjects. At 3 months following Engensis, this improvement was observed in 25% of subjects. Muscle strength was stable for the first 3 months following Engensis administration and then steadily declined in both upper and lower limbs at subsequent months.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically definite or probable Amyotrophic Lateral Sclerosis or laboratory-supported probable Amyotrophic Lateral Sclerosis as defined in the revised El Escorial/Airlie House diagnostic criteria
2. The site of onset of Amyotrophic Lateral Sclerosis symptoms is a limb and experiencing symptoms of lower motor dysfunction (e.g., weakness, atrophy, cramps, poor circulation, etc.) with upper motor neuron symptoms (e.g., weakness, brisk reflexes, spasticity)
3. Onset of Amyotrophic Lateral Sclerosis symptoms ≤ 4 years
4. Slow Vital Capacity ≥ 50% of predicted value at Screening
5. Not taking riluzole, or on a stable dose (defined as no noted toxicities) for at least 30 days prior to Screening and throughout the study
6. Not taking edaravone or on a maintenance cycle for at least 30 days prior to Screening and throughout the study
7. For females of childbearing potential, a negative urine pregnancy test at Screening and on Day 0
8. Male Participants and their female partners must agree to use double-barrier contraception during the study or provide proof of postmenopausal state (minimum 1 year) or surgical sterility
9. Male Participants must not donate sperm during the study
10. Female Participants must be nonpregnant, nonlactating, and either postmenopausal for at least 1 year, or surgically sterile for at least 3 months, or agree to use double-barrier contraception from 28 days prior to randomization (Day 0) and/or their last confirmed menstrual period prior to study randomization (whichever is longer) until the end of the study
11. Capable of complying and willing to comply with the requirements and restrictions in the informed consent form and this protocol
12. Willing to forgo new experimental Amyotrophic Lateral Sclerosis treatments for at least 6 months following randomization

Exclusion Criteria:

1. Progressive or degenerative neurological disorder such as Alzheimer's disease, Parkinson's disease, vascular dementia, multiple sclerosis, and other neurological or vascular disorders felt by the Investigator to preclude participation
2. Requires tracheotomy ventilation or noninvasive ventilation related to bulbar function
3. Evidence by physical examination, history, or laboratory evaluation of significant concomitant disease with a life expectancy of < 6 months at Screening
4. International Normalized Ratio values >2.0
5. Platelet count <100,000/µL
6. Inflammatory disorder of the blood vessels (inflammatory angiopathy or vasculitis, such as Buerger's disease)
7. Active infection (chronic infection or severe active infection that may compromise the Participant's wellbeing or participation in the study in the Investigator's judgment)
8. Chronic inflammatory disease (e.g., Crohn's disease, rheumatoid arthritis)
9. Positive human immunodeficiency virus or human T-cell lymphotrophic virus I/II test at Screening
10. Active acute or chronic hepatitis B
11. Active hepatitis C
12. Immunosuppression due to underlying disease (e.g., rheumatoid arthritis, systemic lupus erythematosus) or to currently receiving immunosuppressive drugs, (e.g., chemotherapy, corticosteroids) or to radiation therapy
13. Stroke or myocardial infarction within 3 months prior to Screening
14. Active deep vein thrombosis
15. Recent history (< 3 years) or presence of cancer except basal cell carcinoma or squamous cell carcinoma of the skin that was excised and has shown no evidence of recurrence for at least 1 year
16. Major psychiatric disorder diagnosed in the past 6 months that has not been stabilized or in the Investigator's opinion would not allow the patient to participate in the scheduled procedures
17. Use of an investigational drug for the treatment of Amyotrophic Lateral Sclerosis in the past 30 days or 5 half-lives (if available), whichever is longer, or previous participation in a clinical study with Engensis
18. Stem cell administration for investigational treatment of Amyotrophic Lateral Sclerosis or other conditions in the 6 months prior to Screening

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-03-09 (Actual); Primary Completion 2022-07-11 (Actual); Study Completion 2024-07-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (4):
  - St. Joseph's Hospital and Medical Center, Barrows Neurological Institute, Phoenix, Arizona
  - Northwestern University, Chicago, Illinois
  - Johns Hopkins University Department of Neurology, Baltimore, Maryland
  - Austin Neuromuscular Center, Austin, Texas
- Hanyang University Medical Center, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Engensis | Placebo
Started | 12 | 6
Completed | 10 | 4
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Engensis | Placebo | Total
Number analyzed (Participants) | 12 | 6 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 6 | 18
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (14.2) | 52.2 (8.45) | 48.1 (12.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 10 | 4 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 6 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 4 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 5 | 2 | 7
  United States | 7 | 4 | 11

OUTCOME MEASURES:

1. Primary Outcome: Safety of Intramuscular Injections of Engensis in Participants With Amyotrophic Lateral Sclerosis Compared to Placebo
Description: Incidence of treatment-emergent adverse events in more than or equal to 10% of subjects, and treatment-emergent serious adverse events after injections, injection site reactions, and clinically significant laboratory values for Engensis compared to Placebo.
Time Frame: From the Day 0 Visit to the Day 180 Visit
Population: Treatment-Emergent Adverse Events in ≥10% of Subjects Overall by System Organ Class and Preferred Term (Safety Analysis Population)
Measure: Count of Participants; unit: Participants
Arm/Group | Engensis | Placebo
Number analyzed (Participants) | 12 | 6
Participants
  Injection Site bruising | 4 | 3
  Pyrexia | 3 | 1
  Injection site pain | 2 | 1
  Asthenia | 0 | 2
  Fatigue | 1 | 1
  Arthralgia | 2 | 0
  Muscle spasms | 1 | 1
  Musculoskeletal stiffness | 2 | 0
  Back pain | 2 | 0
  Joint range of motion decreased | 1 | 1
  Myalgia | 0 | 2
  Muscle contractions involuntary | 2 | 1
  Dysarthria | 1 | 1
  Headache | 1 | 1
  Cough | 3 | 1
  Rhinorrhoea | 2 | 1
  Diarrhoea | 2 | 0
  Nausea | 1 | 1
  COVID-19 | 5 | 1
  Insomnia | 1 | 1
  Hypertension | 1 | 1

2. Other Pre Specified Outcome: Changes in Muscle Function Following Engensis Injections Compared to Placebo
Description: Change from Baseline (Day 0) in total mean Revised Amyotrophic Lateral Sclerosis Function Rating scores, subscores for Fine and Gross Motor Functions and Bulbar Function, and slope of the total score.
  The Revised Amyotrophic Lateral Sclerosis Function Rating scores includes twelve questions that ask the physician to rate his/her impression of the patient's level of functional impairment in performing one of twelve common tasks e.g., climbing stairs). Each task is rated on a five-point scale from 0 = can't do, to 4 = normal ability. Individual item scores are summed to produce a reported score of between 0 = worst and 48 = best. The Revised Amyotrophic Lateral Sclerosis Function Rating scores was conducted at Screening, pre-dose on Days 0, 60, and 120, and on Days 30, 84, 144, and 180.
Time Frame: Day 0 to Day 180
Population: Revised Amyotrophic Lateral Sclerosis Function Rating scores - Change from Baseline to Day 180 (ITT Population)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Engensis | Placebo
Number analyzed (Participants) | 12 | 6
score on a scale | -5.9 (4.2) | -4.2 (4.76)

3. Other Pre Specified Outcome: Evaluation of Muscle Strength Changes Following Engensis Injections Compared to Placebo - Hand-Held Dynamometry
Description: As assessed bilaterally by Hand-Held Dynamometry in muscles in the upper and lower extremities.
  Muscle Strength as Measured by Handheld Dynamometry (lbs.) and Change from Baseline to Day 180 by Muscle Group (ITT Population)
Time Frame: Day 0 to Day 180
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Pounds (lbs.)
Arm/Group | Engensis | Placebo
Number analyzed (Participants) | 12 | 6
Pounds (lbs.)
  Shoulder Flexion, left | -6.48 (8.317) | -3.33 (1.552)
  Shoulder Flexion, right | -7.608 (9.2493) | -2.100 (4.4234)
  Elbow Flexion, left | -10.562 (12.7571) | -3.250 (4.4004)
  Elbow Flexion, right | -10.68 (11.813) | -1.68 (3.174)
  Elbow Extension, left | -6.424 (11.0173) | 2.350 (1.1590)
  Elbow Extension, right | -6.83 (8.925) | -1.08 (5.171)
  Wrist Extension, left | -7.162 (7.8940) | 4.943 (8.5556)
  Wrist Extension, right | -6.53 (10.081) | -2.18 (4.350)
  First Dorsal Interosseous, left | -0.712 (1.2620) | -0.150 (0.3000)
  First Dorsal Interosseous, right | -0.808 (1.0350) | -0.050 (0.1000)
  Abductor Pollicus Brevis, left | -2.188 (2.7008) | 0.200 (0.4000)
  Abductor Pollicus Brevis, right | -2.174 (4.2892) | 0.050 (0.1000)
  Abductor Digiti Minimi, left | -0.17 (1.122) | 0.00 (0.000)
  Abductor Digiti Minimi, right | -1.028 (1.1762) | 0.00 (0.0000)
  Hip Flexion, left | -14.82 (23.235) | 0.15 (23.742)
  Hip Flexion, right | -13.12 (18.239) | -1.88 (20.747)
  Knee Flexion, left | -14.018 (19.2911) | -1.575 (6.2809)
  Knee Flexion, right | -12.64 (11.764) | -1.73 (5.904)
  Knee Extension, left | -14.966 (10.2662) | -1.725 (4.2366)
  Knee Extension, right | -13.022 (6.5484) | 0.125 (5.9690)
  Ankle Dorsiflexion, left | -13.28 (18.262) | -3.80 (3.586)
  Ankle Dorsiflexion, right | -14.30 (15.165) | -4.03 (4.800)

4. Other Pre Specified Outcome: Evaluation of Muscle Strength Changes Following Engensis Injections Compared to Placebo - Accurate Test of Limb Isometric Strength
Description: As assessed bilaterally by the Accurate Test of Limb Isometric Strength where available. Accurate Test of Limb Isometric Strength - Muscle strength values for each muscle group and change from Baseline were presented, neither descriptive statistics presented by visit and treatment group.
Time Frame: Day 0 to Day 180
Population: The Accurate Test of Limb Isometric Strength was not performed on any subject due to sites not being trained or were unable to conduct the procedure.
Arm/Group | Engensis | Placebo
Number analyzed (Participants) | 0 | 0

5. Other Pre Specified Outcome: Evaluation of Quality of Life Improvement Following Engensis Injections Compared to Placebo - Exploratory Outcome
Description: The Amyotrophic Lateral Sclerosis Assessment Questionnaire has 40 items (ALSAQ-40), and is a standardized Quality of Life assessment.
  The Participant completes the 40 questions in the ALSAQ-40 with 5 categories: Physical Mobility, Activities of Daily Living and Independence, Eating and Drinking, Communication, and Emotional Reactions. Each question has 5 responses to select from: 0-Never (Best Case), 1-Rarely, 2-Sometime, 3-Often, and 4-Always (Worst Case).
  Note for each question there is a Minimum of 0 (Best), to the Maximum 4 (Worst). Decreasing scores indicates improvement of symptoms.
  The Total ALSAQ-40 scores are per Category as percentages of 100% maximum. Each Category percentage is summed for the Intent-to-treat Population.
  The Change from Baseline is displayed in the Table. ALSAQ-40 was completed at the pre-dose visit (Day 0), and at the Day 84 and Day 180 visits.
  The Total Change From Baseline is calculated for the Day 84 visit, and the Day 180 visit.
Time Frame: Day 0 to Day 84, and Day 0 to 180
Population: Amyotrophic Lateral Sclerosis Assessment Questionnaire. Percent Change from Baseline (ITT Population) for Engensis and Placebo.
Measure: Mean (Standard Deviation); unit: percentage of Change from Baseline
Arm/Group | Engensis | Placebo
Number analyzed (Participants) | 12 | 6
percentage of Change from Baseline
  Day 84 - Physical Mobility | 1.88 (20.255) | -1.5 (5.755)
  Day 180 - Physical Mobility | 13.44 (24.014) | 11.88 (17.366)
  Day 84 - Activities of Daily Living/Independence | 10.31 (9.396) | 0.50 (8.178)
  Day 180 - Activities of Daily Living/Independence | 15.94 (17.369) | 11.25 (12.332)
  Day 84 - Eating and Drinking | 8.34 (12.596) | 11.66 (21.732)
  Day 180 - Eating and Drinking | 17.73 (18.623) | 14.58 (21.886)
  Day 84 - Communication | 11.15 (24.334) | 7.14 (13.363)
  Day 180 - Communication | 24.56 (27.690) | 11.60 (25.977)
  Day 84 - Emotional Functioning | 7.81 (24.401) | 6.00 (6.755)
  Day 180 - Emotional Functioning | 20.00 (21.423) | 11.25 (11.087)

6. Other Pre Specified Outcome: Evaluation of Patient Reported Outcome Improvement Following Engensis Injections Compared to Placebo
Description: The subject's impression of change after treatment was measured with the Patient Global Impression of Change questionnaire through use of the electronic Patient Reported Outcome . This questionnaire measures the subject's perception of how treatment has affected their level of activity, symptoms, emotions, and overall quality of life.
  Each descriptor is ranked on an increasing improvement scale; where 1 = No change (or condition has got worse), 2=Almost the same, hardly any change at all, 3=A little better, but no noticeable change, 4=Somewhat better, but the change has not made any real difference, 5=Moderately better, and a slight but noticeable change, 6=Better, and a definite improvement that has made a real and worthwhile difference, and 7 = A great deal better, and a considerable improvement that has made all the difference.
  The test was self-administered on Days 84 and 180.
Time Frame: Day 84 and Day 180 (End of Study or Early Termination)
Population: Patient Global Impression of Change - ITT Population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Engensis | Placebo
Number analyzed (Participants) | 12 | 6
score on a scale
  Day 84: number analyzed (Participants) | 8 | 5
  Day 84 | 3.1 (1.81) | 4.6 (0.89)
  End of Study / Early Term- Day 180: number analyzed (Participants) | 8 | 4
  End of Study / Early Term- Day 180 | 2.9 (1.46) | 4.0 (2.00)

7. Other Pre Specified Outcome: Evaluation of Clinical Reported Outcome Improvement Following Engensis Injections Compared to Placebo
Description: The Clinical Global Impression of Change is a validated instrument completed by observers as an assessment of Quality of Life. The Clinical Global Impression of Change is an 8-point scale with scores ranging from Marked Improvement, Moderate Improvement, Minimal Improvement, Slight Improvement, and Unchanged (or Worse), along with an efficacy index with questions in a matrix for therapeutic effect and side effects.The test was completed on Days 84 and 180/ Early Termination.
Time Frame: Day 84 to Day 180
Population: Clinical Global Impression of Change - ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Engensis | Placebo
Number analyzed (Participants) | 12 | 6
Participants
  Day 84 - Minimally improved | 2 | 3
  Day 84 - Minimally worse | 5 | 1
  Day 84 - No change | 3 | 2
  End Study/Early term- Minimally improved | 0 | 1
  End Study/Early term- Minimally worse | 4 | 0
  End Study/Early term- Much worse | 2 | 1
  End Study/Early term- No change | 4 | 2

8. Other Pre Specified Outcome: To Determine Effects of Engensis on Respiratory Function Compared to Placebo - Slow Vital Capacity
Description: Slow vital capacity is a pulmonary function test that quantifies the volume of air that can be slowly exhaled after slow maximum inhalation, and was to be measured at Screening, pre-dose on Days 60 and 120, and on Days 30, 84, 144, and 180.
Time Frame: Day 0 to Day 180
Population: Slow Vital Capacity Percent Change from Baseline by Visit (ITT Population)
Measure: Mean (Standard Deviation); unit: percentage of Change from Baseline
Arm/Group | Engensis | Placebo
Number analyzed (Participants) | 12 | 6
percentage of Change from Baseline
  Day 30 | -3.31 (4.191) | 2.53 (7.501)
  Day 60 (pre-dose) | -6.50 (9.439) | -3.90 (9.173)
  Day 84 | -6.50 (11.808) | -2.3 (9.182)
  Day 120 (pre-dose) | -12.76 (13.363) | -8.84 (12.916)
  Day 144 | -13.46 (17.605) | -9.04 (15.925)
  Day 180 | -17.80 (17.308) | -1.75 (10.046)

9. Other Pre Specified Outcome: To Determine Effects of Engensis on Respiratory Function Compared to Placebo - Tracheostomy
Description: Total Participants that experienced Tracheostomy during the study in the Intent-to-treat population.
Time Frame: Day 0 to Day 180
Population: Participants that Experienced Tracheostomy during the study - ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Engensis | Placebo
Number analyzed (Participants) | 12 | 6
Participants | 0 | 0

10. Other Pre Specified Outcome: To Determine Effects of Engensis on Survival Compared to Placebo - Deaths
Description: Participants that died during the study, for all causes including Treatment Emergent Adverse Events, or Treatment Emergent Serious Adverse Events, leading to study discontinuation, or study drug withdrawal in any subject.
Time Frame: Day 0 to Day 180
Population: Time to All-Cause Death - ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Engensis | Placebo
Number analyzed (Participants) | 12 | 6
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From Day 0 to Day 180 or Early Termination
Description: Treatment Emergent Adverse Events by System Organ Class and Preferred Term Safety Analysis Population
Arm/Group | Engensis | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/6
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/6
Other Adverse Events (participants affected / at risk) | 10/12 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Engensis (N=12) | Placebo (N=6)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Engensis (N=12) | Placebo (N=6)
Injection site bruising (General disorders) | 4 (7) | 3 (9)
Pyrexia (General disorders) | 3 (3) | 1 (1)
Injection site pain (General disorders) | 2 (13) | 1 (1)
Asthenia (General disorders) | 0 (0) | 2 (4)
Fatigue (General disorders) | 1 (1) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Muscle contractions involuntary (Nervous system disorders) | 2 (3) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (2) | 1 (1)
Headache (Nervous system disorders) | 1 (2) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
COVID-19 (Infections and infestations) | 5 (5) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-01-20): https://cdn.clinicaltrials.gov/large-docs/25/NCT04632225/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-05): https://cdn.clinicaltrials.gov/large-docs/25/NCT04632225/SAP_001.pdf